CLINICAL TRIAL: NCT03177525
Title: Parent Training to Enhance Social Success for Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Grace Gengoux, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41867
Record Dates: First submitted 2017-06-01; First posted 2017-06-06 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Autism Spectrum Disorder
Keywords: parent training; social skills
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social SUCCESS (Experimental)
  Interventions: Behavioral: Social SUCCESS
- Wait List (Other)
  Interventions: Behavioral: Wait List

INTERVENTIONS:
Behavioral: Social SUCCESS — Social SUCCESS will run for 12 weeks, with up to 5 children with ASD per group. Parents will attend didactic group sessions focused on motivating children with ASD to initiate to peers (90 min weekly) and will attend a portion of the existing 90 min social group to practice applying these strategies with their children and peer volunteers. Parent training will utilize the manual "Improving Socialization in Individuals with Autism".
  Arms: Social SUCCESS
Behavioral: Wait List — Participants assigned to the Wait List will continue stable community treatments for 12 weeks and will be provided an intervention similar to Social SUCCESS upon completion of all post measures.
  Arms: Wait List

SUMMARY:
Children with autism spectrum disorder (ASD) exhibit characteristic deficits in social initiation and there are no empirically validated treatments specifically for this core deficit. While parent training is known to be a critical intervention component, few social skills programs involve parents. This study will capitalize on an existing social skills group already established at the community agency Abilities United, with the goal of enhancing the program's effectiveness by adding a parent component. Specifically, the proposed study will investigate whether a novel parent mediated social skills program (Social SUCCESS), which provides parent training in conjunction with a social skills group intervention, will result in more frequent initiations during play with typically developing peers. Participants will include 50 children with ASD age 4:0 to 6:11 years. Children will be randomly assigned to either Social SUCCESS (N=25) or waiting list (N=25). Treatment will be provided for 8 weeks during a weekly 120-minute social skills group at Abilities United. The study will evaluate the effects of Social SUCCESS on areas of core social deficit including frequency of peer initiations using parent ratings, observational measures, standardized questionnaires, and a social eye tracking task. Outcomes will be compared to a waiting list control group. Findings will be disseminated through presentations and publications to aid clinicians in providing more effective social skills treatment for children with ASD and to enhance the scientific knowledge-base related to evidence-based social skills treatments. This research designed with the goal of stimulating additional scientific inquiry in the area of treatment for core social deficits in ASD and will provide a strong foundation for larger scale grants to study motivation-based interventions to improve social functioning.

ELIGIBILITY:
Inclusion Criteria:

* child aged 4.0 to 6.11 years
* child diagnosed with ASD (Autism Diagnostic Observation Schedule; ADOS-2)
* child without intellectual disability (Stanford Binet Intelligence Scales; SB-5)
* parent able to consistently participate in parent training sessions and complete study measures

Exclusion Criteria:

* child with other severe psychiatric disorder
* child with known genetic condition (e.g., Fragile X, Retts)
* child with unstable medical condition (e.g., active seizures)

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale Rating from Baseline to Week 12 | Baseline, Week 12
  Parent rating on a Visual Analog Scale (VAS) of the child's frequency of initiation will be compared between Baseline and Week 12 to evaluate change

SECONDARY OUTCOMES:
Change in frequency of child initiations | Baseline, Week 12
  Based on behavioral coding of peer play videos by a blind rater using established operational definitions, change between baseline and week 12 in frequency of child initiations will be compared between groups
Change in parent fidelity of implementation | Baseline, Week 12
  Changes in prompting and reinforcement of social initiations between baseline and week 12 scored from video of parent-child interaction by trained raters will be compared between groups
Social Responsiveness Scale, Second Edition | Baseline, Week 12, 3-month Follow-up
  Social Responsiveness Scale, Second Edition, Parent Report Form
Social Skills Improvement System | Baseline, Week 12, 3-month Follow-up
  Social Skills Improvement System Parent Report Form

CONTACTS AND LOCATIONS:
Overall Officials: Grace W Gengoux, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No